CLINICAL TRIAL: NCT05724784
Title: Development and Feasibility Testing of a Suicide Prevention Intervention for Sexual and Gender Minority Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Candice Biernesser, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22120062
Record Dates: First submitted 2023-01-27; First posted 2023-02-13 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Psychological Distress; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: The study design is an open trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Flourish (Experimental): Participants will be onboarded to Flourish by a research study clinician, following which they will receive a text messaging program for 4 weeks as well as an accompanying resources website.
  Interventions: Behavioral: Flourish

INTERVENTIONS:
Behavioral: Flourish — Flourish is a text messaging program that aims to improve coping following cyberbullying and reduce suicide risk among youth.

SUMMARY:
This study aims to develop and test a brief, digital, suicide prevention intervention for sexual and gender minority (SGM) youth who have experienced cyberbullying. Leading up to this phase, the study team completed two prior study aims, focused on identifying perspectives of SGM youth's regarding their experiences with cyberbullying and priorities for an intervention, and a phase in which SGM youth codesigned the study's intervention with the study team. This resulted in the development of study's intervention, Flourish, which leverages a text messaging-based chatbot to reduce suicide risk following cyberbullying among SGM youth through improving distress tolerance, motivation for help-seeking, and social problem-solving.

Current Study Aim:

Conduct an open trial to assess the feasibility and acceptability of Flourish among cyberbullied SGM youth, ages 12-17 (N=10).

Hypotheses:

Feasibility will be evidenced by recruitment/retention rates > 80% and use of Flourish among > 70% of SGM youth.

At follow-up, adolescents will report improved problem-solving capacity, distress tolerance, and motivation for help-seeking and reduced psychological distress and suicidal ideation compared to baseline.

DETAILED DESCRIPTION:
FLOURISH:

Flourish is a chatbot that will aim to improve adolescents' capacity to cope following cyberbullying and reduce their suicidal risk. The duration of Flourish is 4 weeks. Flourish is designed to be self-paced with branching logic, aiming to provide the right type of support at the right time youth need it. Therefore, the frequency with which youth interact with Flourish will differ from person to person. However, participants are expected to interact with Flourish no less than 2-3 times per week.

Onboarding. Prior to initiating Flourish, adolescents and their caregivers will participate in a session of approximately 30 minutes with a study clinician in which they will onboard to Flourish. During onboarding, the clinician will orient the adolescent to Flourish and load information onto Flourish that will be available to the adolescent throughout their use of the intervention. This will include personal crisis contacts, such as trusted adults and crisis hotlines they could contact in the event of a crisis, as well as contacts for people they could reach out to for support or distraction outside of a crisis situation, such as a close friend or a family member. Adolescents will additionally enter information to personalize their experience with Flourish, such as entering preferences for coping skills that work best for them. During the onboarding process, caregivers will be provided with resources to respond to cyberbullying s as well as information on their child's personal crisis resources.

Launch. The research team will administer brief questionnaires to adolescents 2-3 times per week during the 4-week intervention period that assess positive/supportive and negative/bullying interactions on social media. If adolescents indicate negative interactions, Flourish will automatically launch. If adolescents indicate supportive interactions (or no interactions), they will be given the option to launch Flourish to practice their coping skills, so they are prepared to respond to future cyberbullying events.

Resource Website:

Participants receiving Flourish will also have access to an accompanying website. The website will not collect or store any private information from the participant, and the participant will not interact with the website. It is a publicly available website that provides a list of resources participants may use, if needed. For example, this will include SGM mental health organizations and organizations that provide education, support, and advocacy for youth who have experienced cyberbullying.

Treatment Targets:

To reduce psychological distress and suicidal ideation, Flourish will deploy distress tolerance skills and utilize principles of problem-solving therapy and motivational interviewing.

Problem-Solving. Problem-solving therapy (PST) is a brief cognitive-behavioral intervention that aims to improve coping with stressful life events. PST has shown efficacy in reducing suicide risk among youth and has been successfully delivered in a self-guided online format. Flourish will target: problem identification by aiding youth in appraising the threat of the cyberbullying event they experienced and their socioemotional consequences, generation of potential solutions based on available resources for response, and decision-making through considering barriers and facilitators to putting solutions into action.

Motivation. Motivational Interviewing (MI) is a patient-centered approach that provides a framework for enhancing intrinsic motivation for change that has shown efficacy for improving help-seeking among youth at suicidal risk and has been used in digital mental health interventions. Flourish will incorporate the spirit of MI through its clinical style (i.e., collaborative, empowering language) and MI techniques through responses that are affirming, reflections to demonstrate the chatbot is listening, and offer simple summaries to evoke a change mindset. Flourish will engage strategies to support self-efficacy by focusing on confidence in help-seeking. Through a library of messages, refined to assure fidelity with MI principles, Flourish will elicit thoughts about seeking help following cyberbullying, assess readiness for behavior change through rulers that assess importance and confidence in change, and make a plan for help-seeking. Youth will be offered individualized feedback through stories of SGM adolescents' help-seeking experiences. Developed by writers in partnership with SGM youth, stories will target key motivational barriers to help-seeking following cyberbullying identified in the investigators' pilot data: trust, confidentiality, fear of negative appraisal, and disbelief that help will be effective. Stories will be tailored, i.e., offering examples for youth of differing ages, genders, and identities, and will consider experiences specific to SGM youth of color.

Distress Tolerance. Flourish will be designed to support adolescents' tolerance of distress in recognition that sustained distress experiences contribute to suicidal ideation and interfere with adaptive problem-solving. Flourish will lead youth in monitoring distress levels and respond with a coping skills library that leverages existing online content, focusing on distraction and self-soothing (e.g., guided meditation, breathing exercises, and savoring positive memories).

ELIGIBILITY:
Inclusion Criteria:

* self-reported SGM identity
* English-speaking
* access to a phone or device to complete the study's intervention
* past-month history of cyberbullying or online discrimination, assessed by the cybervictimization subscale of the traditional and cyberbullying victimization and perpetration scale or a discrimination measure developed as part of the Adolescent Brain and Cognitive Development (ABCD) study
* lifetime history of suicidal ideation or behavior (assessed by the Ask Suicide Screen)

Exclusion Criteria:

* intellectual challenges, low literacy levels, or other conditions that might inhibit adolescents' ability to effectively engage with Flourish (reported by parents and, if needed, confirmed through the age-appropriate Wechsler Intelligence scale)
* acuity levels suggesting need for a higher level of care (e.g., inpatient hospitalization) or referral for emergency services

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rates of eligible participants | Assessed upon recruitment to the study
  Feasibility will be measured through recruitment rates of eligible participants, using a cut-off score of 80% for desirable recruitment rates.
Retention rates of eligible participants | Assessed upon completion of the Week 12 study visits
  Feasibility will be measured through retention rates of eligible participants, using a cut-off score of 80% for desirable retention rates across the 12-week study period.
Level of intervention usage | Assessed upon completion of the 4-week intervention period
  Usage of the intervention will be assessed by engagement with the text messaging intervention one or more times during the study period. A cut-off score of 70% of youth using the intervention one or more times will be used as a minimum requirement for acceptable usage.

SECONDARY OUTCOMES:
Change in psychological distress from baseline to 4 weeks | Assessed at the baseline and Week 4 follow-up assessment visits.
  Psychological distress will be measured by the Kessler 6-item psychological distress scale (K6). Total scale scores range from 0 to 24 with higher values indicating higher levels of distress and lower values indicating lower distress.
Change in psychological distress from baseline to 4 weeks | Assessed at the Week 12 follow-up assessment visits.
  Psychological distress will be measured by the Kessler 6-item psychological distress scale. Total scale scores range from 0 to 24, higher values indicating higher levels of distress and lower values indicating lower distress.
Change in severity of suicidal ideation and behavior from baseline to 4 weeks | Assessed at baseline and Week 4 follow-up assessment visits.
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Change in severity of suicidal ideation and behavior from baseline to 12 weeks | Assessed at baseline and Week 12 follow-up assessment visits.
  Severity of suicidal ideation and behavior will be measured with the C-SSRS, an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Change in suicidal ideation from baseline to 4 weeks | Assessed at the baseline and Week 4 assessment visits.
  Self-reported suicidal ideation will be measured with the Suicidal Ideation Questionnaire (SIQ). The SIQ has a total score of 0 to 90. Higher scores are indicative of frequent suicidal ideation, and lower scores indicative of infrequent ideation.
Change in suicidal ideation from baseline to 12 weeks | Assessed at the baseline and Week 12 Follow-up assessment visits.
  Self-reported suicidal ideation will be measured with the Suicidal Ideation Questionnaire. The SIQ has a total score of 0 to 90. Higher scores are indicative of frequent suicidal ideation, and lower scores indicative of infrequent ideation.

OTHER OUTCOMES:
Change in distress tolerance from baseline to 4 weeks | Assessed at the baseline and Week 4 assessment visits
  Distress tolerance will be measured by the Distress Tolerance Scale. The total score for this scale ranges from 15 to 75 with higher scores indicating higher levels of distress tolerance and lower scores indicating lower distress tolerance.
Change in distress tolerance from baseline to 12 weeks | Assessed at the baseline and Week 12 assessment visit.
  Distress tolerance will be measured by the Distress Tolerance Scale. The total score for this scale ranges from 15 to 75 with higher scores indicating higher levels of distress tolerance and lower scores indicating lower distress tolerance.
Change in motivation for help-seeking from baseline to 4 weeks | Assessed at the baseline and Week 4assessment visits.
  Motivation for help-seeking will be measured by Readiness, Importance, and Confidence rulers. This includes three rulers assessing readiness, importance, and confidence in help-seeking following cyberbullying. Scores for each ruler range from 0 (not at all ready) to 10 (very ready).
Change in motivation for help-seeking from baseline to 12 weeks | Assessed at the baseline and Week 12 follow-up assessment visits.
  Motivation for help-seeking will be measured by Readiness, Importance, and Confidence rulers. This includes three rulers assessing readiness, importance, and confidence in help-seeking following cyberbullying. Scores for each ruler range from 0 (not at all ready) to 10 (very ready).
Change in social problem-solving from baseline to 4 weeks | Assessed at baseline and Week 4 assessment visits.
  Social problem-solving will be measured by the revised, short version of the Social Problem-Solving Inventory. This scale has a total score from 0 to 100 with higher scores indicating more effective problem-solving and lower scores representing a less effective problem-solving.
Change in social problem-solving from baseline to 12 weeks | Assessed at the baseline and Week 12 assessment visits.
  Social problem-solving will be measured by the revised, short version of the Social Problem-Solving Inventory. This scale has a total score from 0 to 100 with higher scores indicating more effective problem-solving and lower scores representing a less effective problem-solving.

CONTACTS AND LOCATIONS:
Overall Officials: Candice L Biernesser, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from enrolled participants may be shared with investigators within and outside of the University of Pittsburgh and University of Pittsburgh Medical Center for the purpose of studying cyberbullying or suicide risk among SGM adolescents.
Supporting Information: Study Protocol
Time Frame: These data will be released following acceptance of the project's main outcomes manuscript.
Access Criteria: Data requests may be sent to the PI for review, who will provide data to interested and qualified investigators.